CLINICAL TRIAL: NCT02296424
Title: β-SPECIFIC 4 Patients: Study of Pediatric EffiCacy and Safety wIth FIrst-line Use of Canakinumab An Open-label Canakinumab (ACZ885) Dose Reduction or Dose Interval Prolongation Efficacy and Safety Study in Patients With Systemic Juvenile Idiopathic Arthritis (SJIA)
Brief Title: ß-SPECIFIC 4 Patients: Study of Pediatric EffiCacy and Safety wIth FIrst-line Use of Canakinumab
Acronym: ß-SPECIFIC 4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CACZ885G2306; 2013-004867-29 (EudraCT Number)
Record Dates: First submitted 2014-10-10; First posted 2014-11-20 (Estimated); Results first posted 2019-07-09 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-06

CONDITIONS: Systemic Juvenile Idiopathic Arthritis (SJIA)
Keywords: Juvenile Rheumatoid arthritis (JRA) chronic; systemic inflammatory disorder; painful joints; inflammation of the synovial membrane; auto-immune rheumatoid disease; reactive rheumatoid arthritis; Systemic Juvenile Rheumatoid arthritis (SJRA)
MeSH Terms: conditions — Arthritis, Juvenile; Bronchiolitis Obliterans Syndrome; Arthralgia; Rheumatoid Arthritis, Systemic Juvenile | interventions — canakinumab

STUDY DESIGN:
Intervention Model Description: A two-part open-label study that collected long-term efficacy, safety, and tolerability data from SJIA patients receiving canakinumab treatment who had inactive disease at the last visit in Study CACZ885G2301E1 (Cohort 1), and from SJIA patients who were canakinumab treatment-naïve and had active disease at the time of screening for this study (Cohort 2)
Masking Description: No blinding was required in this open-label study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Canakinumab Dose Reduction (Experimental): All patients received canakinumab 4mg/kg (300 mg max) every 4 weeks in Part I of the study. Patients eligible for Part II of the study were randomized to one of two treatment arms. This is Treatment Arm 1 in Part II of the study: Canakinumab was administered at a reduced dose (2 mg/kg every 4 weeks). If the patient continued to maintain inactive disease for 24 additional weeks, canakinumab was administered at 1mg/kg every 4 weeks. If the patient continued to maintain inactive disease for another 24 additional weeks, canakinumab treatment was discontinued.
  Interventions: Drug: ACZ885 150 mg (Canakinumab)
- Canakinumab Dose Interval Prolongation (Experimental): All participants received canakinumab 4mg/kg (300 mg max) every 4 weeks in Part I of the study. Patients eligible for Part II of the study were randomized to one of two treatment arms. This is Treatment Arm 2 in Part II of the study: Canakinumab dose interval was prolonged to a regimen of 4mg/kg every 8 weeks. If the patient continued to be stable with inactive disease for 24 additional weeks, canakinumab dose interval was prolonged to a regimen of 4mg/kg every 12 weeks. If the patient was clinically stable with inactive disease for another 24 additional weeks, canakinumab treatment was discontinued.
  Interventions: Drug: ACZ885 150 mg (Canakinumab)

INTERVENTIONS:
Drug: ACZ885 150 mg (Canakinumab) — Active canakinumab in individual 2 mL glass vials, each containing 150 mg canakinumab liquid in vial.
  Other Names: ACZ885 150 mg

SUMMARY:
The purpose of this study was to evaluate the efficacy observed with canakinumab dose reduction in a subgroup of patients in the extension study CACZ885G2301E1.

DETAILED DESCRIPTION:
This two-part open-label study was to assess 2 different canakinumab taper regimens in patients with clinical remission (inactive disease for at least 24 continuous weeks) on canakinumab treatment without concomitant corticosteroids (CS) or methotrexate (MTX). The study was also to collect long term safety and tolerability data on SJIA patients treated with canakinumab.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1:

• Patients who are receiving canakinumab treatment (4 mg/kg every 4 weeks) for Systemic Juvenile Idiopathic Arthritis (SJIA) and have inactive disease at the last visit in Study CACZ885G2301E1

Cohort 2:

* Confirmed diagnosis of SJIA as per International League Against Rheumatism (ILAR) definition that must have occurred at least 2 months prior to enrollment with an onset of disease < 16 years of age.
* Active SJIA defined as having 2 or more of the following:
* Documented spiking, intermittent fever (body temperature > 38°C) for at least 1 day within 1 week before first canakinumab dose;
* At least 2 joints with active arthritis
* C-reactive protein (CRP) > 30 mg/L (normal range < 10 mg/L)
* Rash due to SJIA
* Serositis
* Lymphadenopathy
* Hepatosplenomegaly
* Negative TB screen (QuantiFERON or, if required by local guidelines, Purified Protein Derivative).

Exclusion Criteria:

* With active or recurrent bacterial, fungal or viral infection at the time of enrollment, including patients with evidence of Human Immunodeficiency Virus (HIV) infection, Hepatitis B and Hepatitis C infection.
* With underlying metabolic, renal, hepatic, infectious or gastrointestinal conditions which in the opinion of the investigator immunocompromises the patient and /or places the patient at unacceptable risk for participation.
* With neutropenia (absolute neutrophil count < 1500/mm3) at screening.

Ages: 2 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 182 (Actual)
Dates: Start 2014-11-17 (Actual); Primary Completion 2016-10-14 (Actual); Study Completion 2017-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (45):
- United States (2):
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Columbus, Ohio
- Novartis Investigative Site, Vienna, Austria
- Belgium (3):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Laken
  - Novartis Investigative Site, Leuven
- Brazil (3):
  - Novartis Investigative Site, Curitiba, Paraná
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, São Paulo, São Paulo
- Canada (2):
  - Novartis Investigative Site, Vancouver, British Colombia
  - Novartis Investigative Site, Toronto, Ontario
- France (3):
  - Novartis Investigative Site, Bron
  - Novartis Investigative Site, Le Kremlin-Bicêtre
  - Novartis Investigative Site, Paris
- Germany (7):
  - Novartis Investigative Site, Sankt Augustin, North Rhine-Westphalia
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Giessen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Tübingen
- Novartis Investigative Site, Budapest, Hungary
- Israel (5):
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Kfar Saba
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Ramat Gan
- Italy (5):
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Napoli
- Novartis Investigative Site, Utrecht, Netherlands
- Novartis Investigative Site, Warsaw, Poland
- Russia (2):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
- Spain (4):
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Esplugues de Llobregat, Barcelona
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Stockholm, Sweden
- Turkey (Türkiye) (4):
  - Novartis Investigative Site, Istanbul, TUR
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Quartier P, Alexeeva E, Constantin T, Chasnyk V, Wulffraat N, Palmblad K, Wouters C, I Brunner H, Marzan K, Schneider R, Horneff G, Martini A, Anton J, Wei X, Slade A, Ruperto N, Abrams K; Paediatric Rheumatology International Trials Organisation and the Pediatric Rheumatology Collaborative Study Group. Tapering Canakinumab Monotherapy in Patients With Systemic Juvenile Idiopathic Arthritis in Clinical Remission: Results From a Phase IIIb/IV Open-Label, Randomized Study. Arthritis Rheumatol. 2021 Feb;73(2):336-346. doi: 10.1002/art.41488. Epub 2020 Dec 11. PMID 32783351

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 182 enrolled but 16 qualified immediately for Part II & were randomized while 166 continued in Part I & were treated with canakinumab 4 mg/kg every 4 weeks until study end unless they discontinued, or until they qualified for Part II. Of these, 40 discontinued. Most frequent reason was lack of efficacy
Pre-assignment Details: 75 patients (Cohort 1: 56 and Cohort 2: 20) qualified for Study Part II and were randomized to receive canakinumab at either a reduced dose (n=38) or a prolonged dose interval (n=37)
Groups:
- Cohort 1: Participants from study CACZ885G2301E1, aged ≥ 2 to < 20 years at the time of the patient's first dose of canakinumab, who at the time of evaluation for participation in CACZ885G2306 were being treated with canakinumab 4mg/kg and had inactive disease
- PART 1: Cohort 2: Participants who at screening were aged ≥ 2 to < 20 years, had active SJIA (as per protocol), and were canakinumab treatment-naïve
- Dose Reduction; Dose Interval Prolongation: canakinumab 4 mg/kg every 4 weeks until study end unless discontinuation occurred, or until they qualified & entered Part II
Period: Part 1
Arm/Group | Cohort 1 | PART 1: Cohort 2 | Dose Reduction | Dose Interval Prolongation
Started | 84 (16 patients immediately went into Part II) | 98 | 0 | 0
Completed | 61 | 65 | 0 | 0
Not Completed | 23 | 33 | 0 | 0
Not completed — New therapy for study indication | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 0
Not completed — Study terminated by sponsor | 0 | 1 | 0 | 0
Not completed — Adverse Event | 2 | 11 | 0 | 0
Not completed — Lack of Efficacy | 5 | 17 | 0 | 0
Not completed — 16 directly started part II | 16 | 0 | 0 | 0
Period: Part 2
Arm/Group | Cohort 1 | PART 1: Cohort 2 | Dose Reduction | Dose Interval Prolongation
Started | 0 | 0 | 38 | 37
Completed | 0 | 0 | 35 | 37
Not Completed | 0 | 0 | 3 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Set
  All patients who received at least one dose of study drug in Cohort 1 (resp. in Cohort 2) and had at least one post-treatment safety assessment in Part I before the canakinumab dose reduction/interval prolongation part. Of note, the statement that a patient had no adverse events (AE) also constituted a safety assessment.
Groups:
- Cohort 2: Dose interval prologation All participants received canakinumab 4mg/kg (300 mg max) every 4 weeks in Part I of this study
  All participants in Part II of this study came from Part 1, So only Part 1 is shown here in Baseline Characteristics
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 68 | 98 | 166
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Safety Set
  Years
    Age (years) | 11.8 (4.53) | 8.3 (4.20) | 9.7 (4.66)
Age, Customized [Number; unit: participants] — Population: Safety Set
  participants
    >=2 - <4 years: number analyzed (Participants) | 1 | 14 | 15
    >=2 - <4 years | 1 | 14 | 15
    >=4 - <6 years: number analyzed (Participants) | 6 | 17 | 23
    >=4 - <6 years | 6 | 17 | 23
    >=6 - <12 years: number analyzed (Participants) | 24 | 42 | 66
    >=6 - <12 years | 24 | 42 | 66
    >=12 - <20 years: number analyzed (Participants) | 34 | 25 | 59
    >=12 - <20 years | 34 | 25 | 59
    >=20 years: number analyzed (Participants) | 3 | 0 | 3
    >=20 years | 3 |  | 3
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Safety Set
  Participants
    Female | 34 | 42 | 76
    Male | 34 | 56 | 90
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 66 | 81 | 147
  More than one race | 1 | 12 | 13
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants in Clinical Remission on Canakinumab Who Are Able to Remain at an Initial Reduced Canakinumab Dose or Prolonged Canakinumab Dose Interval.
Description: The primary efficacy variable for Part II was the proportion of patients in clinical remission on canakinumab 4 mg/kg (+/- concomitant NSAID only) who were able to remain on a reduced dose or on prolonged dose interval for at least 24 consecutive weeks. As the primary objective was to show statistically significance in at least one of canakinumab treatment arms (reduced dose and prolonged dose interval arms) in Part II then the Type I error rate 5% was controlled and split to 2.5%. Clinical remission per protocol is defined as the maintenance of inactive disease for at least 6 months (24consecutive weeks) while on therapy. The primary analysis considered both inactive disease status and the patient dose step duration.
  In the event the inactive disease status was missing, yet the patient remained at the same dose level through the next visit with the same disease status, it was concluded that inactive disease was maintained during this time period and was carried forward.
Time Frame: baseline to 24 weeks
Population: Full Analysis Set
Measure: Number; unit: particiapants
Groups:
- Canakinumab Dose Reduction: Cohort 1 In total, 75 patients (Cohort 1: 56 and Cohort 2: 20) qualified for Study Part II and were randomized to receive canakinumab at either a reduced dose (n=38) or a prolonged dose interval (n=37)
- Canakinumab Dose Interval Prolongation: Cohort 2 In total, 75 patients (Cohort 1: 56 and Cohort 2: 20) qualified for Study Part II and were randomized to receive canakinumab at either a reduced dose (n=38) or a prolonged dose interval (n=37)
Arm/Group | Canakinumab Dose Reduction | Canakinumab Dose Interval Prolongation
Number analyzed (Participants) | 38 | 37
particiapants
  Able to remain on dose: number analyzed (Participants) | 11 | 6
  Able to remain on dose | 27 | 31
  Not able to remain on dose | 11 | 6
Statistical Analysis 1: Comparison: Canakinumab Dose Reduction vs Canakinumab Dose Interval Prolongation; Test type: Equivalence — nominal 2.5% two-sided significance level was expected to have 90% powe to detect a difference between the Null Hypothesis proportion of patients who remain at their dose level; p = 0.0001, exact binomial test

2. Secondary Outcome: Number and Percentage of Patients With Adverse Events as a Measure of Long-term Safety and Tolerability of Canakinumab - PART 1
Description: AEs, Deaths, other serious adverse events or discontinuations due to AE, Part I (Safety set)
Time Frame: During study parts I and II. The estimated study duration is not more than 216 weeks (with an average expected duration of 108 weeks).
Population: Safety Set
Measure: Number; unit: number of participants
Groups:
- Canakinumab Dose Interval Prolongation: Cohort 2 All patients received canakinumab 4mg/kg (300 mg max) every 4 weeks in Part I of the study. Patients eligible for Part II of the study were randomized to one of two treatment arms. This is Treatment Arm 2 in Part II of the study: Canakinumab dose interval was prolonged to a regimen of 4mg/kg every 8 weeks. If the patient continued to be stable with inactive disease for 24 additional weeks, canakinumab dose interval was prolonged to a regimen of 4mg/kg every 12 weeks. If the patient was clinically stable with inactive disease for another 24 additional weeks, canakinumab treatment was discontinued.
Arm/Group | Canakinumab Dose Reduction | Canakinumab Dose Interval Prolongation
Number analyzed (Participants) | 68 | 98
number of participants
  Number of patients with at least one AE | 57 | 91
  Number of patients with death | 0 | 0
  Number of patients with at least one SAE | 10 | 23

3. Secondary Outcome: Number and Percentage of Patients With Adverse Events as a Measure of Long-term Safety and Tolerability of Canakinumab - PART 2
Description: AEs, Deaths, other serious adverse events or discontinuations due to AE, Part II (Safety set)
Time Frame: During study parts I and II, estimated study duration was not more than 216 weeks (with an average duration of 108 weeks).
Population: Safety Set
Measure: Number; unit: number of participants
Arm/Group | Canakinumab Dose Reduction | Canakinumab Dose Interval Prolongation
Number analyzed (Participants) | 38 | 37
number of participants
  Number of patients with at least one AE | 38 | 34
  Number of patients with death | 0 | 0
  Number of patients with at least one SAE | 4 | 1

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All AEs reported in this record are from date of First Patient First Treatment until Last Patient Last Visit) up to estimated study duration of not more than 216 weeks (with an average duration of 108 weeks)
Description: Arms/Groups are combined because a threshold of 5% indicates that all Other (Not Including Serious) Adverse Events with a frequency greater than 5% within at least one arm or comparison group are reported.
Groups:
- Part I: Part I
- Part II@Dose Reduction: Part II@Dose reduction
- Part II@Dose Interval@Prolongation: Part II@Dose interval@prolongation
Arm/Group | Part I | Part II@Dose Reduction | Part II@Dose Interval@Prolongation
All-Cause Mortality (participants affected / at risk) | 0/166 | 0/38 | 0/37
Serious Adverse Events (participants affected / at risk) | 33/166 | 4/38 | 1/37
Other Adverse Events (participants affected / at risk) | 140/166 | 38/38 | 34/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part I (N=166) | Part II@Dose Reduction (N=38) | Part II@Dose Interval@Prolongation (N=37)
Histiocytosis haematophagic (Blood and lymphatic system disorders) | 3 | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Pericarditis (Cardiac disorders) | 2 | 0 | 0
Eye swelling (Eye disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0
Atypical pneumonia (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 2 | 0 | 0
Infectious mononucleosis (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Otitis media (Infections and infestations) | 1 | 1 | 0
Otitis media acute (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Viral infection (Infections and infestations) | 2 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Juvenile idiopathic arthritis (Musculoskeletal and connective tissue disorders) | 8 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Still's disease (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Idiopathic intracranial hypertension (Nervous system disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Alveolar proteinosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Lichen planus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash scarlatiniform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part I (N=166) | Part II@Dose Reduction (N=38) | Part II@Dose Interval@Prolongation (N=37)
Lymphadenopathy (Blood and lymphatic system disorders) | 10 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 13 | 5 | 6
Abdominal pain upper (Gastrointestinal disorders) | 14 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 18 | 4 | 2
Nausea (Gastrointestinal disorders) | 11 | 3 | 3
Vomiting (Gastrointestinal disorders) | 17 | 3 | 0
Injection site reaction (General disorders) | 13 | 2 | 1
Pyrexia (General disorders) | 33 | 9 | 12
Bronchitis (Infections and infestations) | 9 | 5 | 2
Gastroenteritis (Infections and infestations) | 12 | 3 | 5
Influenza (Infections and infestations) | 16 | 5 | 3
Nasopharyngitis (Infections and infestations) | 34 | 10 | 10
Pharyngitis (Infections and infestations) | 19 | 2 | 6
Respiratory tract infection (Infections and infestations) | 16 | 3 | 1
Rhinitis (Infections and infestations) | 23 | 4 | 4
Tonsillitis (Infections and infestations) | 8 | 3 | 5
Upper respiratory tract infection (Infections and infestations) | 23 | 8 | 6
Viral infection (Infections and infestations) | 9 | 5 | 3
Iron deficiency (Metabolism and nutrition disorders) | 10 | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 25 | 8 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 3 | 3
Juvenile idiopathic arthritis (Musculoskeletal and connective tissue disorders) | 21 | 6 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 3 | 7
Headache (Nervous system disorders) | 26 | 5 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 23 | 9 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 17 | 6 | 3
Eczema (Skin and subcutaneous tissue disorders) | 15 | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 16 | 3 | 5
Urticaria (Skin and subcutaneous tissue disorders) | 9 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 7 | 0 | 2
Conjunctivitis allergic (Eye disorders) | 2 | 1 | 2
Constipation (Gastrointestinal disorders) | 3 | 4 | 2
Gastritis (Gastrointestinal disorders) | 1 | 2 | 1
Odynophagia (Gastrointestinal disorders) | 0 | 2 | 0
Toothache (Gastrointestinal disorders) | 3 | 2 | 0
Fatigue (General disorders) | 7 | 2 | 0
Oedema peripheral (General disorders) | 0 | 0 | 2
Conjunctivitis (Infections and infestations) | 3 | 2 | 4
Cystitis (Infections and infestations) | 2 | 2 | 2
Ear infection (Infections and infestations) | 2 | 0 | 2
Gastroenteritis viral (Infections and infestations) | 4 | 0 | 2
Hordeolum (Infections and infestations) | 3 | 2 | 1
Otitis externa (Infections and infestations) | 1 | 2 | 0
Otitis media (Infections and infestations) | 3 | 3 | 0
Otitis media acute (Infections and infestations) | 4 | 1 | 2
Pharyngotonsillitis (Infections and infestations) | 1 | 2 | 0
Urinary tract infection (Infections and infestations) | 4 | 3 | 0
Varicella (Infections and infestations) | 5 | 2 | 2
Contusion (Injury, poisoning and procedural complications) | 4 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 3
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 2
Ligament sprain (Injury, poisoning and procedural complications) | 5 | 0 | 2
Blood creatine phosphokinase increased (Investigations) | 2 | 3 | 1
Lipase increased (Investigations) | 3 | 2 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0 | 2
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 1 | 2 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 2 | 2 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 4 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.